CLINICAL TRIAL: NCT00686530
Title: Comparison of Abnormal Cortical Development in Brain Malformations on Postmortem Imaging With Autopsy
Status: Withdrawn | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Susan Blaser, Neuro Radiologist, The Hospital for Sick Children
Other Study IDs: 1000011050
Record Dates: First submitted 2008-05-23; First posted 2008-05-30 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2008-05

CONDITIONS: Brain Malformation
Keywords: Fetal Death; Magnetic Resonance Imaging; Autopsy; Telencephalon; Pyramidal Tracts
MeSH Terms: conditions — Fetal Death | interventions — Magnetic Resonance Spectroscopy; Autopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Macroscopic examination of the fetus will be performed initially follwed by organ removal for tissue fixation for a period of two weeks.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: MR Imaging; Procedure: Autopsy

INTERVENTIONS:
Procedure: MR Imaging — Postmortem MR will be included as part of the autopsy examination in cases of suspected brain malformations. Imaging will be done using 1.5T GE CV/I MRI magnet. The specimen is scanned, following fixation, using an 8-channel head coil or 8-channel knee coil, depending on the size of the brain. Structural postmortem MR will include spin-echo T1, axial SPGR, and T2 imaging in three planes. Diffusion tensor imaging will be performed in the coronal plane.
Procedure: Autopsy — Autopsy will be performed according to accepted standards, based on clinical indications. Macroscopic examination of the fetus will be performed initially , followed by organ removal for tissue fixation for a period of two weeks.

SUMMARY:
Examination of the fetal brain at autopsy is technically challenging because of marked fragility of the brain tissue. Studies have found postmortem fetal MR to be particularly useful in examining gross structural abnormalities in fetal brain and spine. We have recently included postmortem MR as part of the radiological studies for fetal autopsy workup. Using the same MR data, the development of normal layering of the brain, also called laminar organization, can also be assessed. This laminar organization of the brain is often disturbed in congenital malformations. Our aim is to study the disturbance in laminar organization of the postmortem brain with MR, using structural MR and a type of MR sequence called diffusion tensor imaging, which is well suited for assessing the organization of the developing brain. The postmortem MR findings will be compared with gold standard of histopathology. This will help us understand the abnormal development of gray and white matter in brain malformations. Knowledge gained from studying the abnormal laminar organization in brain malformations will serve as a reference for future studies of fetal brain malformations in-utero using MRI.

DETAILED DESCRIPTION:
1. Autopsy will be performed at Mount Sinai Hospital according to accepted current standards, based on clinical indications. Macroscopic examination of the fetus will be performed initially, followed by organ removal for tissue fixation for a period of two weeks. The brain is then scanned with MRI at the Hospital for Sick Children. The brain is transported in an air-tight container containing 10% formalin and sealed with paraffin lined tape. All brains will be anonymised and coded with a number prior to MRI examination. Following MR imaging, the tissue will be examined, sampled and reported in the usual fashion at Mount Sinai Hospital.
2. Postmortem MR will be included as part of the autopsy examination in cases of suspected brain malformations. Postmortem MR will be performed at the Hospital for Sick Children due to availability of expertise in postmortem neuroimaging and imaging will be done using 1.5T GE CV/I MRI magnet (General Electric, Milwaukee, WI). Postmortem MR will be performed following dissection and tissue fixation to avoid any unnecessary delay in tissue fixation. The specimen will be scanned in an air-tight container containing formalin 10%, sealed with paraffin lined tape. Structural postmortem MR will include coronal spin-echo T1 (TR=517msec, TE=10msec, FOV=18cm, slice thickness=20-30mm, matrix=320x256), axial SPGR (TR=23msec, TE=8msec, FOV=18cm, slice thickness=1.1mm, matrix=256x256) and T2 imaging in three planes (TR=4115msec, TE=115msec, FOV=16cm, slice thickness=20-30mm, matrix=320x256). Diffusion tensor imaging (TR=8300msec, TE=99msec, FOV=180mm, slice thickness=2-3mm, b=700mm/sec2, NEX=8, matrix=128x128, 25 directions) will be performed in the coronal plane to match the histological sections of brain tissue in autopsy.
3. Analysis. The laminar organization of the fetal cerebrum on structural MR and diffusion tensor imaging will be evaluated. In particular, the germinal matrix, intermediate zone, subplate and cortex will be assessed. This will be compared with the gold standard of histopathology. The presence or absence of corticospinal tracts will also be assessed and compared with macroscopic examination and histological sections.
4. Statistical analysis. The sensitivity, specificity and accuracy of postmortem MR, both structural and diffusion tensor imaging, as compared to the gold standard of autopsy in assessing the abnormal laminar organization of fetal cerebrum will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* suspected antenatal diagnosis of brain malformation who will undergo autopsy and MRI to further assess the malformations
* above 18 weeks gestation

Exclusion Criteria:

* significant autolysis of tissue specimens prior to tissue fixation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40 fetal post mortem brains, with suspected diagnosis of brain malformation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Estimated); Study Completion 2010-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaser, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario